CLINICAL TRIAL: NCT07016997
Title: A Phase I Study to Assess the Safety, Tolerability and Biomarker Profiles of CBA-1535, Recombinant Protein Tribody in Patients With Previously Treated Advanced Solid Tumors.
Brief Title: A Phase I, First in Human Study of CBA-1535, T Cell Engager(5T4/CD3/5T4) in Patients With Advanced Solid Tumors.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chiome Bioscience Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1535-001; jRCT2031210708 (Other Grant/Funding Number: Japan Registry of Clinical Trials)
Record Dates: First submitted 2025-04-07; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumors; Refractory Cancer
Keywords: CBA-1535; 5T4; CD3; T cell Engager; Trophoblast Glycoprotein; Tribody; solid tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: CBA-1535 (single agent therapy) (Experimental): Patients will receive CBA-1535 as weekly IV infusion at escalated doses on Day 1, 8 and 15 of each 21-day cycle.
  Interventions: Drug: CBA-1535
- Part 2: CBA-1535+Pembrolizumab (Experimental): Patients will receive CBA-1535 as weekly IV infusion at escalated doses on Day 1, 8 and 15 , and Pembrolizumab as Q3W IV infusion at fix dose on Day 1 of each 21-day cycle.
  Interventions: Drug: CBA-1535+Pembrolizumab

INTERVENTIONS:
Drug: CBA-1535 — Dosing is increased from 0.1 µg/body until DLT or disease progression occurs.
  Arms: Part 1: CBA-1535 (single agent therapy)
Drug: CBA-1535+Pembrolizumab — Drug：CBA-1535 First Dosing will be determined by Part 1. And dosing will be increased until DLT or disease progression occurs.
  Drug：Pembrolizumab 200 mg/body
  Arms: Part 2: CBA-1535+Pembrolizumab

SUMMARY:
This is a First in Human muticenter, non-randomized, open-label Phase I dose-escalation study of CBA-1535.

The study will have 2 parts (Part 1 and Part 2). Part 1 is the dose-escalation cohorts of CBA-1535 single agent theapy. Part 2 is the dose-escalation cohorts of CBA-1535 in combination with Pembrlizumab.

This study will evaluate the safety, tolerability, PK, biomarker profiles and preliminary efficacy of CBA-1535.

DETAILED DESCRIPTION:
To evaluate safety and efficacy of CBA-1535 in the following two parts in a stepwise manner:

Part 1

- In Part 1, the primary objective is to evaluate the safety and tolerability of CBA-1535 in patients with solid tumors where no standard treatment is available, or who are intolerant to or non-responders to standard treatments.

Additionally, the PK, biomarker profiles, and preliminary efficacy will be evaluated. The initial dose for Part 2 will also be determined.

Part 2

- In Part 2, The primary objective is to evaluate the safety and tolerability of CBA-1535 in combination with pembrolizumab in patients with solid tumor where no standard treatment is available, or who are intolerable or non-responder to the standard treatment. Additionally, the PK, biomarker profiles, preliminary efficacy will be evaluated. The recommended Phase 2 dose (R2PD) will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients who provide voluntary written informed consent to participate in the study
* ECOG performance status: <= 1
* Patients with 3 months or longer life expectancy
* Patients with solid tumors for whom no standard therapy is available or who are refractory to or intolerant of standard therapy

Exclusion Criteria:

* Patients who received other investigational drug or antibody drugs, including immune checkpoint inhibitor within 28 days prior to enrollment
* Patients who received anti-cancer drug within 14 days prior to enrollment
* Patients with previous or suspected hypersensitivity to protein preparations such as therapeutic antibodies (Chinese hamster ovary cell-derived drugs) or any component of the study drug

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | Up to 21 days in Cycle 1
  DLTs are assessed according to CTCAE v.5.0 during the first cycle (21 days).
Adverse event | Up to approximately 24 months
  An adverse event is any untoward or unintended sign, symptom, or disease in a subject administered an investigational product, regardless of whether or not it is related to the investigational product.

SECONDARY OUTCOMES:
Serum CBA-1535 concentration | From Day 1 to Day 22
  Blood samples are collected to assess the serum concentration of CBA-1535.
Efficacy in previously treated advanced solid Tumors. | Up to approximately 24 months.
  Efficacy evaluation based on RECIST v.1.1 is performed by CT or MRI scan or others.

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Shizuoka Cancer Center, Nagaizumicho, Shizuoka
  - National Cancer Center Hospital, Chuo-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No